CLINICAL TRIAL: NCT07318181
Title: Fostering Ukraine's Capacity in the Delivery and Research of Innovative Evidence-based PTSD Treatment
Brief Title: Building Ukraine's Strength in PTSD Treatment and Research
Acronym: Lux4UA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luxembourg (Other)
Collaborators: National Psychological Association of Ukraine (Unknown); Veteran Mental Health and Rehabilitation Center 'Forest Glade' Ministry of Health of Ukraine (Unknown); Quresta, Inc. (Unknown)
Responsible Party: Principal Investigator, Viktoriia GORBUNOVA, Sc.D, Research Scientist, University of Luxembourg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-AGR-7624-00; 19403469/LuxAid-Bridges (Other Grant/Funding Number: The Luxembourg National Research Fund)
Record Dates: First submitted 2025-11-28; First posted 2026-01-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder; Post Traumatic Stress Disorder PTSD; Post-Traumatic Stress Disorder, PTSD
Keywords: Post Traumatic Stress Disorder; RTM; RTM Protocol; PTSD; trauma therapy; traumatic memories; memory reconsolidation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Eye Movement Desensitization Reprocessing; Sertraline

STUDY DESIGN:
Intervention Model Description: Participants are assigned by randomised allocation to RTM or TAU using a parallel-group design. Randomisation follows CONSORT guidance for parallel-group trials and employs a covariate-adaptive randomisation technique. To enhance the external validity of the findings, all the interventions are to be explored among three different settings of mental health care accustomed to Ukraine: mental health hospital care (inpatient and outpatient care for veterans) and psychotherapeutic practice (for civil trauma survivors).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: RTM Protocol (Experimental): RTM Protocol - A manualised, algorithmic, imagery-based procedure delivered in 3-5 sessions (~90 minutes each) on consecutive days or with at least one sleep cycle between sessions.
  Interventions: Behavioral: Reconsolidation of Traumatic Memories Protocol
- Arm B: Treatment-as-Usual (TAU) (Active Comparator): Treatment-as-Usual (TAU) - Evidence-based care per routine practice (TF-CBT or EMDR or Selective Serotonin Reuptake Inhibitors) following organisational and professional standards in Ukraine. All interventions in this arm are approved in Ukraine (see Ministry of Health of Ukraine. (2024). Unifikovanyi klinichnyi protokol. Hostra reaktsiia na stres. Posttravmatychnyi stresovyi rozlad. Porushennia adaptatsii [Clinical protocol for acute stress reactions, post-traumatic stress disorder (PTSD), and adaptation disorders] (Order No. 1265). Ministry of Health of Ukraine. https://www.dec.gov.ua/wp-content/uploads/2024/07/1265_19072024_ykpmd_ptsr_dod.pdf)
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy; Behavioral: Eye Movement Desensitization and Reprocessing; Drug: Selective Serotonin Reuptake Inhibitors: Paroxetine, Sertraline

INTERVENTIONS:
Behavioral: Reconsolidation of Traumatic Memories Protocol — The protocol as a structured, mandatory-to-administrate 89-step procedure consists of three main phases: Pre-treatment, Treatment, and Retelling of the Trauma Event. Aside from establishing therapeutic rapport and framing the work, one of the key tasks in the Pre-treatment phase is the Visual Formats Practice. This involves specially organised exercises that help a person engage in imaginative activities with neutral events, preparing them to do similar work addressing trauma in the subsequent steps. The Treatment phase implies leading a person through three types of Visual Formats, specific techniques used to help clients visualise the trauma story in a way that minimises the distress of recalling. The Retelling of the Trauma Event phase intersperses with Visual Formats and serves to assess of so-called subjective distress throughout persons' retelling of traumatic events.
  Other Names: RTM Protocol
  Arms: Arm A: RTM Protocol
Behavioral: Trauma-Focused Cognitive Behavioral Therapy — TF-CBT is designed to help individuals process and recover from traumatic experiences by integrating trauma-sensitive strategies with cognitive-behavioral techniques. It combines psychoeducation, relaxation strategies, emotional regulation, cognitive restructuring, and the development of a trauma narrative to reduce symptoms of PTSD, anxiety, and depression.
  Other Names: TF-CBT
  Arms: Arm B: Treatment-as-Usual (TAU)
Behavioral: Eye Movement Desensitization and Reprocessing — EMDR is a structured, evidence-based psychotherapy designed to help individuals process and heal from traumatic experiences by using bilateral stimulation, typically guided eye movements, while recalling distressing memories. EMDR does not require detailed discussion of the trauma or homework between sessions.
  Arms: Arm B: Treatment-as-Usual (TAU)
Drug: Selective Serotonin Reuptake Inhibitors: Paroxetine, Sertraline — Paroxetine and Sertraline, both SSRIs, are distinguished in PTSD treatment by their strong evidence base and official FDA approval specifically for this condition. They effectively target core PTSD symptoms such as intrusive thoughts, hyperarousal, and emotional numbing by enhancing serotonin regulation. Compared to other pharmacological options, SSRIs offer superior safety, tolerability, and dosing flexibility, making them suitable for long-term use.
  Arms: Arm B: Treatment-as-Usual (TAU)

SUMMARY:
The Lux4UA project aims to support mental health treatment in Ukraine, especially for those who have experienced traumatic events due to the ongoing conflict and forced displacement. As rates of Post-Traumatic Stress Disorder (PTSD) rise among civilians, military personnel, and refugees, the need for effective trauma care becomes urgent. PTSD is a mental health condition that can develop after experiencing trauma, leading to flashbacks, nightmares, anxiety, and other symptoms that significantly impact daily life.

This project introduces an innovative method called the Reconsolidation of Traumatic Memories (RTM) Protocol, which helps individuals reduce distressing memories and trauma-related symptoms. Unlike traditional therapies, the RTM Protocol aims to quickly alleviate PTSD symptoms without requiring patients to relive or discuss in detail their traumatic experiences, which can sometimes be overwhelming. Instead, it employs carefully guided imaginary exercises to help patients reprocess and feel less emotional distress when recalling traumatic memories. This structured approach can lead to significant improvements in just three to five sessions.

The Lux4UA project brings together mental health professionals and researchers from Ukraine, Luxembourg, and the United States to test how well this treatment works in Ukraine and to understand if it can be easily integrated into the country's mental health system. By studying the RTM Protocol in three main settings-hospital care and outpatient (walk-in) clinics for veterans and therapy practices for civilians-the project will assess the treatment's effectiveness for people with different needs and backgrounds. It will also evaluate how comfortable and satisfied both mental health practitioners and patients are with the treatment.

A key part of the project is training Ukrainian mental health professionals in the RTM Protocol. This training ensures that local mental health professionals are well-prepared to deliver the treatment and support trauma survivors long after the project ends, building a sustainable mental health system in Ukraine. The project will involve careful monitoring of how patients respond to the treatment, paying special attention to their well-being throughout each session.

To evaluate the treatment's success, the project will measure changes in PTSD symptoms, as well as signs of anxiety and depression that often accompany trauma. The project will also assess the RTM Protocol's adaptability to Ukrainian needs, seeing if any modifications are necessary to better suit the local context.

DETAILED DESCRIPTION:
The Lux4UA Project aims to strengthen Ukraine's capacity to deliver and research innovative, evidence-based treatment for post-traumatic stress disorder (PTSD) in the context of ongoing war, displacement, and humanitarian crisis. The project evaluates the effectiveness and feasibility of the Reconsolidation of Traumatic Memories (RTM) Protocol - a short-term, neurobiologically grounded intervention that reduces trauma-related symptoms without requiring patients to retell their traumatic experiences in detail.

The Russian invasion of Ukraine has led to a steep rise in PTSD prevalence. Recent studies show that 30-50% of civilians, 55% of internally displaced persons, and over 60% of refugees present with PTSD symptoms, while combat-related PTSD among military personnel is widespread. The Ukrainian mental health system, although reforming toward community-based care, lacks sufficient evidence-based tools to address this unprecedented demand.

Traditional trauma therapies such as trauma-focused cognitive behavioural therapy (TF-CBT), exposure therapy, and eye movement desensitization and reprocessing (EMDR) are recommended by international guidelines and effective in many settings. However, they require lengthy treatment, demand that patients retell traumatic events, and often show high dropout rates (up to 30%). In contrast, RTM Protocol has demonstrated rapid and lasting reductions in PTSD symptoms, often in three to five sessions, with low dropout rates. Randomized controlled trials in the USA and UK report diagnostic remission in 70-88% of veterans treated, with sustained results up to a year post-treatment. These features make RTM Protocol particularly promising for conflict-affected populations where resources are limited and stigma or retraumatization hinder treatment.

A cornerstone of the project is training 20 Ukrainian mental health professionals in the delivery of the RTM Protocol. Training is conducted by Quresta Inc. (USA) in collaboration with the University of Luxembourg, followed by biweekly supervision and accreditation. This ensures both fidelity to the protocol and sustainability. Trained professionals will continue applying RTM beyond the project, potentially treating many trauma survivors in the years ahead.

Data will be collected, pseudonymized in Ukraine by implementing partners - the Centre of Mental Health and Rehabilitation "Forest Glade" of the Ministry of Health of Ukraine (RCFG) and the National Psychological Association of Ukraine (NPAU), and transferred in fully anonymized, aggregated form to the University of Luxembourg for analysis. Findings will inform humanitarian response policy and sustainable capacity-building for evidence-based PTSD treatment in low-resource, conflict settings.

The RTM Protocol effectiveness study implies a randomized field trial with parallel group design, adhering to CONSORT standards, comparing RTM with treatment-as-usual (Trauma-Focused Cognitive Behavioural Therapy (TF-CBT), Eye Movement Desensitisation and Reprocessing (EMDR), or pharmacotherapy) across three customary clinical settings in Ukraine (hospital in-patient, hospital out-patient, private psychotherapy). The primary outcome is the loss of Post-Traumatic Stress Disorder (PTSD) diagnosis or change in symptoms; secondary outcomes include depression and anxiety at post-treatment, 6-month and 12-month follow-up.

Objective 1: To compare the effectiveness of the RTM Protocol for the treatment of trauma-related mental conditions with other evidence-based trauma-focused therapies (TF-CBT, EMDR and medication).

Objective 2: To investigate the effectiveness of the RTM Protocol for the treatment of trauma-related mental conditions in different settings of mental health (MH) care (in-patient and out-patient hospital care for veterans and private psychotherapy for civilians)

The RTM Protocol and Training feasibility study will evaluate the RTM Protocol's acceptability and adaptability during training and practice through case statistics, satisfaction surveys of MH practitioners and clients, and focus-group interviews with MH practitioners.

Objective 1: To analyze the acceptability of the RTM Protocol among MH professionals and persons with trauma-related MH conditions.

Objective 2: To analyze the adaptability (Usability of the Ukrainian language versions) of the RTM Protocol.

The project addresses ethical issues at every stage:

Professional eligibility: Only licensed clinicians with a minimum of three years' experience in trauma care will be considered for training.

Informed consent: All participants (both clinicians and patients) will provide written informed consent.

Data protection: Data are anonymized, stored securely, and processed according to EU GDPR and Ukrainian legislation.

Patient safety: Clear procedures are in place for managing distress, adverse events, and unexpected findings. Participants may withdraw from or switch to a different treatment at any time.

The Lux4UA project spans 36 months and is structured into four work packages:

1. Project Management and Administration - research protocol development, ethics approval, data management, and coordination.
2. RTM Training and Supervision - recruitment and training of professionals, ongoing supervision and certification.
3. RTM Protocol Effectiveness and Feasibility Evaluation - recruitment of 120 patients, intervention delivery, data collection, and analysis.
4. Dissemination and Communication - publication of findings, conference presentations, and policy recommendations.

By combining research, training, and system integration, the Lux4UA project will not only provide and explore trauma treatment but also lay the foundation for a sustainable, evidence-based mental health infrastructure in Ukraine.

ELIGIBILITY:
Inclusion Criteria:

1. being adults 18-65 years,
2. having a diagnosis of PTSD determined by DSM-5-TR or ICD-11 and/or
3. having PTSD symptoms causing clinically significant distress or impact on social, occupational, or other areas of functioning, as defined by the PTSD Checklist PCL-5,
4. being a resident of Ukraine.

Exclusion Criteria:

1. having any other acute comorbid mental health conditions,
2. receiving any other parallel PTSD treatment,
3. being unable to provide informed consent, having severe cognitive impairment, or being otherwise unlikely to adhere to study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
PTSD symptoms according to the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Data collection will occur at baseline, 1 month after complete treatment application, in 6 months, and in 12 months.
  The PCL-5 is a 20-item self-report measure with scores ranging from 0 to 80, with each item rated on a scale from 0 (Not at all) to 4 (Extremely). Higher scores indicate worse outcomes, reflecting greater severity of PTSD symptoms, while lower scores suggest fewer or less severe symptoms.

SECONDARY OUTCOMES:
Anxiety-related symptoms according to the Generalized Anxiety Disorder-7 (GAD-7) | Data collection will occur at baseline, 1 month after complete treatment application, in 6 months, and in 12 months.
  The GAD-7 is a 7-item self-report measure of anxiety severity, with scores ranging from 0 to 21, where each item is rated from 0 (Not at all) to 3 (Nearly every day). Higher scores indicate worse outcomes, reflecting greater severity of anxiety symptoms, while lower scores suggest fewer or less severe symptoms.
Depression-related symptoms according to the Patient Health Questionnaire-9 (PHQ-9) | Data collection will occur at baseline, 1 month after complete treatment application, in 6 months, and in 12 months.
  The PHQ-9 is a 9-item self-report measure of depression severity, with scores ranging from 0 to 27, where each item is rated from 0 (Not at all) to 3 (Nearly every day). Higher scores indicate worse outcomes, reflecting greater severity of depressive symptoms, while lower scores suggest fewer or less severe symptoms.

OTHER OUTCOMES:
Satisfaction with the therapeutic procedure for clients assessed using an 11-item Likert-scale questionnaire | Up to 24 hours after completion of treatment.
  Satisfaction with the therapeutic procedure will be assessed using an 11-item Likert-scale questionnaire designed for mental health professionals. The questionnaire covers three domains: Process Comfort, Expected and Reached Results, and Changes in Trauma Narrative. Each item is rated from 1 (Strongly disagree) to 5 (Strongly agree), with total scores ranging from 11 to 55. Higher scores indicate greater satisfaction with the treatment process and outcomes.
Satisfaction with the therapeutic procedure for mental health professionals assessed using an 11-item Likert-scale questionnaire | Post-treatment completion (up to 1 week after the last assigned client session).
  Satisfaction with the therapeutic procedure will be assessed using an 11-item Likert-scale questionnaire designed for mental health professionals. The questionnaire covers three domains: Process Comfort, Expected and Reached Results, and Changes in Trauma Narrative. Each item is rated from 1 (Strongly disagree) to 5 (Strongly agree), with total scores ranging from 11 to 55. Higher scores indicate greater satisfaction with the therapeutic process and perceived effectiveness for clients.
Usability of the RTM Protocol assessed using the Intervention Usability Scale | Post-treatment completion (up to 1 week after the last assigned client session).
  Usability of the RTM Protocol will be assessed using the standardized Intervention Usability Scale, which consists of 10 items evaluating perceived ease of use, complexity, integration of components, confidence in use, and need for support. Each item is rated on a 5-point Likert scale (1 = Strongly disagree to 5 = Strongly agree), with total scores ranging from 10 to 50. Higher scores indicate greater usability and confidence in applying the RTM Protocol.
MH professionals' feedback | Post-treatment completion (up to 1 week after the last assigned client session).
  The feedback of MH professionals will also be considered during the focus group analysis. The script previews topics such as the RTM Protocol use features, the RTM Protocol implementation benefits and challenges, the RTM Protocol effects and consequences, the RTM Protocol clients' acceptance and perception, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoriia V Gorbunova, ScD, Principal Investigator — University of Luxembourg
Locations (2):
- Ukraine (2):
  - National Psychological Association of Ukraine, Kyiv
  - Veteran Mental Health and Rehabilitation Center 'Forest Glade' Ministry of Health of Ukraine, Kyiv

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the therapists and research coordinators who will collect data. This decision is based on the high sensitivity of the data, which involves trauma histories and mental health information from children. Even with de-identification, the small sample size and the vulnerability of the population create a risk of re-identification. For these reasons, only anonymised data will be shared with researchers, and only aggregated results will be shared through publications and presentations.

REFERENCES:
- [Result] Gorbunova V, Hampton R. The Reconsolidation of Traumatic Memories Protocol's adjustments to the remote treatment of injured Ukrainian military personnel in hospital settings. Eur J Psychotraumatol. 2025 Dec;16(1):2499410. doi: 10.1080/20008066.2025.2499410. Epub 2025 May 19. PMID 40387497
- [Result] Sturt J, Rogers R, Armour C, Cameron D, De Rijk L, Fiorentino F, Forbes T, Glen C, Grealish A, Kreft J, Meye de Souza I, Spikol E, Tzouvara V, Greenberg N. Reconsolidation of traumatic memories protocol compared to trauma-focussed cognitive behaviour therapy for post-traumatic stress disorder in UK military veterans: a randomised controlled feasibility trial. Pilot Feasibility Stud. 2023 Oct 13;9(1):175. doi: 10.1186/s40814-023-01396-x. PMID 37833734
- [Result] Astill Wright L, Horstmann L, Holmes EA, Bisson JI. Consolidation/reconsolidation therapies for the prevention and treatment of PTSD and re-experiencing: a systematic review and meta-analysis. Transl Psychiatry. 2021 Sep 3;11(1):453. doi: 10.1038/s41398-021-01570-w. PMID 34480016

DOCUMENTS (3):
  • Study Protocol (2025-12-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT07318181/Prot_000.pdf
  • Informed Consent Form: Professionals (2025-12-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT07318181/ICF_002.pdf
  • Informed Consent Form: Clients (2025-12-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT07318181/ICF_001.pdf